CLINICAL TRIAL: NCT07334860
Title: A Two-Period, Open-label, Fixed-Sequence Study to Evaluate the Single-Dose Pharmacokinetics of Two Formulations of MK-1167 in Healthy Participants
Brief Title: A Clinical Trial to Compare Forms of MK-1167 in Healthy People (MK-1167-011)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 1167-011; MK-1167-011 (Other: MSD)
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: MK-1167 Form 2 (Experimental): Participants receive MK-1167 Form 2 orally.
  Interventions: Drug: MK-1167
- Arm 2: MK-1167 Form 1 (Experimental): Participants receive MK-1167 Form 1 orally.
  Interventions: Drug: MK-1167

INTERVENTIONS:
Drug: MK-1167 — Oral administration

SUMMARY:
Researchers are looking for new ways to treat Alzheimer's disease (AD). AD is a brain disease that causes a gradual decline in memory, thinking, and ability to carry out daily tasks. MK-1167 is a study medicine designed to treat symptoms of AD. Before giving a study medicine to people with a health condition, researchers first do studies in healthy people to find a safe dose of the study medicine.

The goals of the trial are to learn:

* What happens to different forms of MK-1167 in a healthy person's body over time
* About the safety of MK-1167 and if people tolerate it

ELIGIBILITY:
Inclusion Criteria:

* Is in good health
* Has a body mass index (BMI) ≥18 and ≤ 32 kg/m^2, inclusive

Exclusion Criteria:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological abnormalities or diseases
* Is a smoker and/or has used nicotine or nicotine-containing products within the past 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-02-04 (Estimated); Primary Completion 2026-05-28 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve from Time 0 to Infinity (AUC0-inf) of MK-1167 | At designated time points (up to approximately 21 days)
  Blood samples will be collected to determine the AUC0-inf of MK-1167.
Maximum Plasma Concentration (Cmax) of MK-1167 | At designated time points (up to approximately 21 days)
  Blood samples will be collected to determine the Cmax of MK-1167.
Area Under the Curve from Time 0 to Last Measurable Concentration (AUC0-last) of MK-1167 | At designated time points (up to approximately 21 days)
  Blood samples will be collected to determine the AUC0-last of MK-1167.

SECONDARY OUTCOMES:
Area Under the Curve from Time 0 to 24 hours (AUC0-24) of MK-1167 | At designated time points (up to approximately 24 hours)
  Blood samples will be collected to determine the AUC0-24 of MK-1167.
Concentration at 24 hours (C24) of MK-1167 | At designated time points (up to approximately 24 hours)
  Blood samples will be collected to determine the C24 of MK-1167.
Time to Maximum Serum Concentration (Tmax) of MK-1167 | At designated time points (up to approximately 21 days)
  Blood samples will be collected to determine the Tmax of MK-1167.
Apparent Terminal Half-life (t1/2) of MK-1167 | At designated time points (up to approximately 21 days)
  Blood samples will be collected to determine the t1/2 of MK-1167.
Apparent Clearance after Nonintravenous Administration (CL/F) of MK-1167 | At designated time points (up to approximately 21 days)
  Blood samples will be collected to determine the CL/F of MK-1167.
Apparent Volume of Distribution during Terminal Phase (Vz/F) of MK-1167 | At designated time points (up to approximately 21 days)
  Blood samples will be collected to determine the Vz/F of MK-1167.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 78 days
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 36 days
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com